CLINICAL TRIAL: NCT00433563
Title: A 2-Arm Randomized Controlled Trial of Concurrent Chemo-Radiotherapy Comparing Twice-Daily and Once-Daily Radiotherapy Schedules in Patients With Limited Stage Small Cell Lung Cancer (SCLC) and Good Performance Status [CONVERT]
Brief Title: Concurrent Once Daily Versus Twice Daily Radiotherapy for Limited Stage Small Cell Lung Cancer
Acronym: CONVERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Cancer Research UK (Other); NCIC Clinical Trials Group (Network); European Organisation for Research and Treatment of Cancer - EORTC (Network); Spanish Lung Cancer Group (Other); Groupe Francais De Pneumo-Cancerologie (Other); Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000531709; CHNT-CONVERT (Other: Christie Hospital NHS Foundation Trust); CHNT-CTAAC-CONVERT-C17052/A815 (Other Grant/Funding Number: Cancer Research UK)
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Once daily radiotherapy (Experimental): Once daily radiotherapy
  Interventions: Radiation: Once daily radiotherapy; Radiation: Twice daily radiotherapy
- Twice daily radiotherapy (Active Comparator): Twice daily radiotherapy
  Interventions: Radiation: Once daily radiotherapy; Radiation: Twice daily radiotherapy

INTERVENTIONS:
Radiation: Once daily radiotherapy — Standard of care chemotherapy (cisplatin/etoposide) + once daily radiotherapy
Radiation: Twice daily radiotherapy — Standard of care chemotherapy (cisplatin/etoposide) + twice daily radiotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known which schedule of radiation therapy is more effective when given together with chemotherapy in treating small cell lung cancer.

PURPOSE: This randomized phase III trial is studying two different schedules of radiation therapy to compare how well they work when given together with cisplatin and etoposide in treating patients with limited stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare overall survival of patients with limited stage small cell lung cancer treated with chemoradiotherapy comprising cisplatin, etoposide, and once vs twice daily radiotherapy.

Secondary

* Compare local progression-free survival of patients treated with these regimens.
* Compare metastasis-free survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare response rates in patients treated with these regimens.
* Compare the cytotoxic dose intensity of these regimens in these patients.
* Compare the dose intensity of two different schedules of radiotherapy in these patients.

OUTLINE: This is a multicenter, randomized, controlled study. Patients are stratified according to participating center, ECOG performance status (0-1 vs 2), and lactic dehydrogenase, sodium, and alkaline phosphatase levels. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cisplatin IV over 2 hours on days 1-3 OR on day 1 only and etoposide IV over 45-90 minutes on days 1-3. Treatment repeats every 21 days for up to 6 courses. During course 2, patients undergo concurrent radiotherapy once daily 5 days a week for 6½ weeks (total of 33 fractions).
* Arm II: Patients receive cisplatin and etoposide as in arm I. During courses 2 and 3, patients undergo concurrent radiotherapy twice daily 5 days a week for 3 weeks (total of 30 fractions).

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Beginning 3-4 weeks after completion of chemoradiotherapy, patients in both arms achieving a complete or partial response with no evidence of brain metastasis undergo prophylactic cranial irradiation once daily 5 days a week for 2 weeks (total of 10 fractions).

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 532 patients will be accrued for this study.

ELIGIBILITY:
Inclusion/exclusion criteria:

* Either sex, age ≥18 years
* Performance status ECOG grade 0-1. Patients with PS 2 whose general condition is explained by obstructive/bulky disease likely to improve after the first cycle of chemotherapy can be included at the discretion of the local investigator. Patients with PS 2 as a result of comorbid conditions will be excluded.
* Histologically or cytologically confirmed SCLC
* No patients with mixed small-cell and non-small-cell histologic features
* No history of previous malignancy in the last 5 years (except non melanomatous skin or in-situ cervix carcinoma). Patients with previous malignancies (except breast cancer) and in remission for at least 5 years can be included.
* Limited stage disease (Veterans Administration Lung Cancer Study Group) ie patients whose disease can be encompassed within a radical radiation portal.
* No pleural or pericardial effusions proven to be malignant
* RT target volume acceptable by the local radiotherapist
* Pulmonary function

  1. FEV1 >1 litre or 40% predicted value
  2. KCO (DLCO/VA) >40%predicted
* Maximum of one of the following adverse biochemical factors:

  1. Serum alkaline phosphatase more than >1.5 times the upper limit of normal (ULN)
  2. Serum sodium < Lower limit of Normal
  3. Serum LDH > ULN
* Normal serum creatinine and calculated creatinine clearance >50 ml/min. If calculated creatinine clearance is <50 ml/mn according to the Cockroft and Gault formula, an EDTA clearance should be performed
* Adequate haematological function

  1. Neutrophils >1.5 x 109/l
  2. Platelets >100 x 109/l
* Adequate liver function: ALT & AST <= 2.5 x ULN
* No other previous or concomitant illness or treatment which in the opinion of the clinician will interfere with the trial treatments or comparisons
* No prior surgical resection of the primary tumour, no prior radiotherapy for lung cancer
* Considered fit to receive any of the trial regimens
* Female patients must satisfy the investigator that they are not pregnant, or are not of child-bearing potential, or are using adequate contraception. Men must also use adequate contraception, as etoposide is clastogenic.
* Patients must not be breastfeeding
* Patient has read the patient information sheet and has signed the consent form.
* Patients available for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2008-04; Primary Completion 2016-02 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | August 2015

SECONDARY OUTCOMES:
Local progression-free survival | August 2015
Metastasis-free survival | August 2015
Toxicity of treatment | August 2015
Cytotoxic dose intensity | August 2015
Radiotherapy dose intensity | August 2015

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Faivre-Finn, MD, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

REFERENCES:
- [Derived] Tay RY, Fernandez-Gutierrez F, Foy V, Burns K, Pierce J, Morris K, Priest L, Tugwood J, Ashcroft L, Lindsay CR, Faivre-Finn C, Dive C, Blackhall F. Prognostic value of circulating tumour cells in limited-stage small-cell lung cancer: analysis of the concurrent once-daily versus twice-daily radiotherapy (CONVERT) randomised controlled trial. Ann Oncol. 2019 Jul 1;30(7):1114-1120. doi: 10.1093/annonc/mdz122. PMID 31020334
- [Derived] Salem A, Mistry H, Hatton M, Locke I, Monnet I, Blackhall F, Faivre-Finn C. Association of Chemoradiotherapy With Outcomes Among Patients With Stage I to II vs Stage III Small Cell Lung Cancer: Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2019 Mar 1;5(3):e185335. doi: 10.1001/jamaoncol.2018.5335. Epub 2019 Mar 14. PMID 30520977
- [Derived] Faivre-Finn C, Snee M, Ashcroft L, Appel W, Barlesi F, Bhatnagar A, Bezjak A, Cardenal F, Fournel P, Harden S, Le Pechoux C, McMenemin R, Mohammed N, O'Brien M, Pantarotto J, Surmont V, Van Meerbeeck JP, Woll PJ, Lorigan P, Blackhall F; CONVERT Study Team. Concurrent once-daily versus twice-daily chemoradiotherapy in patients with limited-stage small-cell lung cancer (CONVERT): an open-label, phase 3, randomised, superiority trial. Lancet Oncol. 2017 Aug;18(8):1116-1125. doi: 10.1016/S1470-2045(17)30318-2. Epub 2017 Jun 20. PMID 28642008
- [Derived] Groom N, Wilson E, Faivre-Finn C. Effect of accurate heart delineation on cardiac dose during the CONVERT trial. Br J Radiol. 2017 May;90(1073):20170036. doi: 10.1259/bjr.20170036. Epub 2017 Mar 31. PMID 28362511
- [Derived] Colaco R, Sheikh H, Lorigan P, Blackhall F, Hulse P, Califano R, Ashcroft L, Taylor P, Thatcher N, Faivre-Finn C. Omitting elective nodal irradiation during thoracic irradiation in limited-stage small cell lung cancer--evidence from a phase II trial. Lung Cancer. 2012 Apr;76(1):72-7. doi: 10.1016/j.lungcan.2011.09.015. Epub 2011 Oct 19. PMID 22014897
- [Derived] Sheikh H, Colaco R, Lorigan P, Blackhall F, Califano R, Ashcroft L, Taylor P, Thatcher N, Faivre-Finn C. Use of G-CSF during concurrent chemotherapy and thoracic radiotherapy in patients with limited-stage small-cell lung cancer safety data from a phase II trial. Lung Cancer. 2011 Oct;74(1):75-9. doi: 10.1016/j.lungcan.2011.01.020. Epub 2011 Feb 26. PMID 21353720